CLINICAL TRIAL: NCT03239574
Title: MightySat - Clinical Performance Comparison Study
Status: Completed | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-18810A
Record Dates: First submitted 2017-08-01; First posted 2017-08-04 (Actual); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- MightySat Test group (Experimental): The subjects will be enrolled into the test group and will receive the MightySat investigational pulse oximeter.
  Interventions: Device: MightySat

INTERVENTIONS:
Device: MightySat — MightySat - investigational pulse oximeter that will be placed on the subject's right index finger for the duration of the study

SUMMARY:
This study compares the performance of respiratory rate from pleth (RRp) measured with MightySat device on healthy subjects.Subjects will be asked to breathe at specific rates ranging from 5 to 30 breaths per minute.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years old
* Physical status of ASA I or II
* Must be able to read and communicate in English
* Has signed all necessary related documents, e.g. written informed consent, confidentiality agreement
* Passed health assessment screening
* Negative pregnancy test for female subjects of child bearing potential

Exclusion Criteria:

* Younger than 18 years old, older than 45 years old
* ASA physical status of III, IV, and V
* Subject has any medical condition which in the judgement of the investigator, renders them inappropriate for participation in the study
* Inability to tolerate sitting still or minimal movement for at least 30 minutes
* Positive pregnancy test for female subjects
* Refusal to take pregnancy test for women of child bearing potential
* Nursing female subjects
* Refusal of male subjects to agree to shave hair off areas where sensors will be applied (neck)
* Excluded at Principal Investigator's discretion

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Clinical Lab, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MightySat Test Group
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MightySat Test Group
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 10
  Asian or Pacific Islander | 3
  Caucasian | 15
  Hispanic | 5
  Middle Eastern | 1
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of RRp Determination
Description: Accuracy will be determined by comparing the noninvasive respiratory rate by pleth (RRp) measurement of the MightySat to the respiratory rate (RR) reference and calculating the arithmetic root mean square error (Arms) value. In order to obtain the Arms value, the RR measurement from the reference is subtracted from the MightySat RRp measurement for a number of samples, the average of this difference is computed as the bias. The standard deviation of the differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the Arms Error value.
Time Frame: approximately 30-40 minutes
Measure: Number; unit: breaths per minute
Arm/Group | MightySat Test Group
Number analyzed (Participants) | 34
breaths per minute | 1.9

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | MightySat Test Group
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT03239574/Prot_SAP_000.pdf